CLINICAL TRIAL: NCT01620606
Title: Parent Training to Address Pediatric Functional Abdominal Pain
Brief Title: Managing Childhood Abdominal Pain
Acronym: MCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of North Carolina (Other); MultiCare Mary Bridge Children's Hospital & Health Center (Other)
Responsible Party: Principal Investigator, Rona Levy, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13744 SCH
Record Dates: First submitted 2012-02-14; First posted 2012-06-15 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Pediatric Abdominal Pain
Keywords: FAP; RAP; Abdominal Pain; IBS
MeSH Terms: conditions — Abdominal Pain | interventions — Cognitive Behavioral Therapy; Educational Status; Palliative Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SLCBT (Experimental): Social Learning and Cognitive Behavioral Therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy & Social Learning
- SLCBT-R (Experimental): Phone-based Social Learning and Cognitive Behavioral Therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy & Social Learning
- ES (Active Comparator): Education and Support
  Interventions: Behavioral: Education and Support

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy & Social Learning — Cognitive Behavioral Therapy & Social Learning
  Arms: SLCBT; SLCBT-R
Behavioral: Education and Support — Education about the GI system, nutrition and food safety
  Arms: ES

SUMMARY:
Functional abdominal pain (FAP) is a common complaint of childhood, associated with considerable health care costs, disruption of normal activity, emotional distress, and long-term health effects. The study will test a treatment approach which, if successful, would substantially change the treatment for FAP and potentially for a wide range of childhood medical problems where parental responses to symptoms contribute to these adverse effects. The study would also provide a model which would be much more accessible than traditional face-to-face therapies to a broader range of families in need than are currently served.

DETAILED DESCRIPTION:
Functional Abdominal Pain (FAP) affects 10 to 15% of children and has significant social, emotional, and financial costs, but no known organic cause and no accepted medical or behavioral treatment. The researchers have conducted studies that provide support for a theoretical model in which cognitive-behavioral and social learning processes (modeling and/or potentially reinforcing responses by parents) may contribute to the maintenance of illness behaviors and functional disability in children with FAP. The researchers subsequently tested a social learning and cognitive-behavioral intervention for parent-child dyads which focused on changing these parent behaviors as well as teaching coping skills to children. Results support the effectiveness of the intervention and the explanatory value of the theory, demonstrating that parental change is a key element in reducing children's symptoms. The proposed study will build on these findings by evaluating a parent-only intervention. Furthermore, our experience and that of other investigators indicates that alternative intervention models are needed for wider accessibility to the intervention for families in need. While a parent-only format is expected to increase accessibility, we will also evaluate the use of a remote telephone intervention.

ELIGIBILITY:
Inclusion Criteria:

* The child is 7 to 12 years old
* The child experienced at least three episodes of unexplained abdominal pain over a three month period which affected the child's activities
* The child lived with the primary caregiver for at least the last 3 months
* The child and the parent agree to the conditions of study participation, including randomization, participation in intervention and follow-up evaluations
* The parent and child comprehend and speak English without assistance

Exclusion Criteria:

* The child has positive physical or laboratory findings which would explain the abdominal pain
* The child has a chronic disease (e.g. Crohn's, ulcerative colitis, pancreatitis, diabetes, epilepsy, etc.)
* The child is lactose intolerant
* The child had major surgery in the past year
* The parent or child has developmental disabilities that require full-time special education or that impair ability to respond to assessment measures

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 316 (Actual)
Dates: Start 2011-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Abdominal Pain Index | Baseline, 1 week post treatment session 3, 3 months post treatment session 3, 6 months post treatment session 3, 12 months post treatment session 3

SECONDARY OUTCOMES:
Adults' Responses to Children's Symptoms | Baseline, 1-3 days post treatment session 1, 1-3 days post treatment session 2,1 week post treatment session 3, 3 months post treatment session 3, 6 months post treatment session 3, 12 months post treatment session 3
Pain Response Inventory | Baseline, 1 week post treatment session 3, 3 months post treatment session 3, 6 months post treatment session 3, 12 months post treatment session 3
Pain Beliefs Questionnaire | Baseline, 1 week post treatment session 3, 3 months post treatment session 3, 6 months post treatment session 3, 12 months post treatment session 3
Pain Catastrophizing Scale | Baseline, 1-3 days post treatment session 1, 1-3 days post treatment session 2,1 week post treatment session 3, 3 months post treatment session 3, 6 months post treatment session 3, 12 months post treatment session 3

CONTACTS AND LOCATIONS:
Overall Officials: Rona L Levy, MSW, MPH, PhD, Principal Investigator — University of Washington; Miranda vanTilburg, PhD, Principal Investigator — University of North Carolina
Locations (3):
- United States (3):
  - University of North Carolina, Chapel Hill, North Carolina
  - Seattle Children's Hospital, Seattle, Washington
  - Mary Bridge Children's Hospital, Tacoma, Washington

REFERENCES:
- [Derived] Levy RL, Langer SL, van Tilburg MAL, Romano JM, Murphy TB, Walker LS, Mancl LA, Claar RL, DuPen MM, Whitehead WE, Abdullah B, Swanson KS, Baker MD, Stoner SA, Christie DL, Feld AD. Brief telephone-delivered cognitive behavioral therapy targeted to parents of children with functional abdominal pain: a randomized controlled trial. Pain. 2017 Apr;158(4):618-628. doi: 10.1097/j.pain.0000000000000800. PMID 28301859